# Virtual Diabetes Specialty Clinic: A Study Evaluating Remote Initiation of Continuous Glucose Monitoring VDiSC Study

# **Statistical Analysis Plan**

Version: 1.0

Version Date: 12/30/2020

Author: Dan Raghinaru

Based on Protocol Version: 2.0

Note: The table shells are included in a separate document.

# **Revision History**

The following table outlines changes made to the Statistical Analysis Plan.

| Version Number | Author | Approver | Effective Date | Study Stage |
|---|---|---|---|---|
| 1.0 | Dan Raghinaru | Peter Calhoun | 12/30/2020 | Study Enrollment |

| Version Number | Revision Description |
|----------------|----------------------|

# **Approvals**

| Role | Digital Signature or Handwritten Signature/Date |
|---|---|
| Author: Dan Raghinaru | |
| Senior Statistician: Peter Calhoun | |
| JCHR Sponsor Representative: Robin Gal | |

# 1 Statistical and Analytical Plans

- 2 This document summarizes the proposed analyses to be performed for the Virtual Diabetes
- 3 Specialty Clinic (VDiSC) study. All analyses are exploratory and additional analyses and
- 4 outcomes not pre-specified here may be performed in the future. The table shells detailing how
- 5 the results will be displayed will be shown in a separate document.

6

1

# 2 Study Overview

7 8

9

The following two tables gives an overview of the VDiSC study.

10 11

# **Table 1. Study Overview**

12

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Title | Virtual Diabetes Specialty Clinic: A Study Evaluating Remote Initiation |
| | of Continuous Glucose Monitoring |
| Précis | This study will assess feasibility and efficacy of establishing a virtual |
| | diabetes clinic with a focus on introduction of CGM technology and |
| | ongoing CGM use to minimize such rate-limiting factors as geography, |
| | cost and access to specialty care |
| Objectives | The objective of this study is to evaluate a virtual diabetes clinic model, |
| | for adults with either T1D or T2D, that supports integration of CGM into |
| | diabetes self-management and use of decision support technology. |
| Study Design | Single-arm prospective longitudinal study |

| • Ag • Di • the • is o use rec inf • Se • Re • Re du rec de vir • Us rec • Ac • Ur • W: Exclusi • Us sys • Cu dia me du • Fe bro • Cu • Ac • Ex use • Kr ide | on Criteria e ≥18 years old agnosis of type 1 diabetes or type 2 diabetes and using insulin rapy (at least 3 injections of insulin per day or insulin pump that compatible with Tidepool software) Multiple daily injection (MDI) for must be willing to use a device provided by the study that ords the injection dosages and/or enter insulin dosing ormation through an app e a healthcare provider at least once a year sident of United States and plan to reside in the U.S. for the ration of the study This requirement is due to virtual clinic license ruirements and U.S. use restrictions for some study software and vices. Not all U.S. states may be eligible for inclusion due to tual clinic license status. e either an Android or iOS smartphone that is compatible with app uirements that are needed for the study cess to a compatible computer with internet derstand written and spoken English lling and able to follow the study procedures as instructed on Criteria e of real-time CGM (including Abbott Libre or integrated pump |
|---|---|
| • Pa stu • Pla du Inc res cli Sample Size The rec Outcomes Efficac <70 mg | inned relocation to a state other than current state of residence ring the study if virtual clinic is not licensed in the new state. Iividuals working routinely in a state other than current state of idence in the next six months are also ineligible if the virtual nic is not licensed in that state. Tuitment target is 300 initiating CGM. Y Outcomes: CGM use; CGM metrics for hypoglycemia (<54 and /dL), hyperglycemia (>180 and >250 mg/dL), time in range (70- |
| 180 mg<br>variatio<br>and dial<br><b>Safety</b> | dL), mean glucose, and glycemic variability (coefficient of n); HbA1c; participant- reported outcomes including psychosocial petes treatment satisfaction questionnaires |
| Participant Duration Study p Protocol Overview/Synopsis Patient Adults: therapy | Outcomes: Severe hypoglycemia, diabetic ketoacidosis, izations, and emergency room visits |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | may be recruited through insurance providers, primary care networks, or health care providers. |
| | Baseline Data Collection Baseline data collected will include demographics, height and weight, socioeconomic status, diabetes history, knowledge of and experience with diabetes devices, medical history and medications, and health-related physical activity. Questionnaires will collect information related to hypoglycemia awareness, treatment satisfaction, and psychosocial issues. Participant contact information will be collected. Contact information for the participant's diabetes healthcare provider will also be collected. |
| | HbA1c Participant will receive fingerstick HbA1c kits that will be sent to a central lab for measurement after enrollment and at 13 weeks, 26 weeks, 39 weeks, and 52 weeks. |
| | Contact between Study Team and Participant Each participant will be assigned to work with virtual clinic team members. Mental health service support options for diabetes-related mental health issues will be discussed as needed. |
| | Virtual clinic team members will check in with participants during study follow up to review CGM data and recommendations related to diabetes management. |
| | CGM Use Participants will use a blinded CGM device for a single sensor wear period prior to CGM initiation. Participants may be asked to use a blinded CGM for an additional sensor wear period(s) if enough CGM data are not available to establish a baseline that can be used as baseline comparator data. Virtual training will include CGM set up, sensor insertion, alerts and alarms, uploading data, and visualizing data. |
| | Changes in Insulin Dosing If the virtual clinic team believes that changes in insulin type or dosing should be considered, they will work with the participant to implement any such changes. Decision support tools, which include use of a mobile application, may be used if available to provide the virtual clinic team with potential recommendations regarding insulin use. |

**Table 2. Schedule of Visits and Procedures** 

| | | | | | | Clinic Training Ph<br>(0-13 Weeks) | | | Extended<br>Virtual Clinic<br>Follow Up<br>Phase | Optional<br>Participant<br>Follow Up |
|---|---|---|---|---|---|---|---|---|---|---|
| | Enrollment | Initial Virtual<br>Clinic Contact | Baseline CGM<br>Data Collection | Training 1<br>(Week 0) | Training 2<br>(Week 1) | Training 3<br>(Week 3) | CGM Follow<br>Up<br>(Weeks 4, 8) | CGM Follow Up<br>(Week 13) | Follow up<br>(>13-26<br>Weeks) | Follow Up<br>(>26-52 Weeks) |
| TARGET WINDOW | | Within 7 Days<br>from<br>Completion of<br>Enrollment<br>Questionnaires | | Day 0 | Day 7-14 | Day 21-28 | | Weeks 12-14 | | |
| ICF • Eligibility Confirmation | x | | | | | | | | X* | X* |
| Baseline Data Collection Contact Information Demographics Medical History Questionnaires | х | | х | | | | | | | |
| Follow-Up Data Collection** | | | | | х | Х | Х | Х | Х | Х |
| HbA1c*** | | | х | | | | | х | Х | х |
| Video Tutorials / Access to<br>Resource Materials | | Examples:<br>CGM Overview<br>Parts of CGM | Examples:<br>HbA1c Sample<br>Collection<br>CGM Setup | Examples:<br>Understanding<br>Your Real-Time<br>Data<br>How to Change<br>Sensor | Examples: How to Upload CGM Data How to View Reports Understanding Your Ambulatory Glucose Profile / Data Patterns | х | x | x | x | |
| Contact with Study Team <sup>†</sup> | | Х | х | CGM Initiation | CGM Data<br>Interpretation | CGM Data<br>Review<br>Goal Setting | Х | Х | Х | |
| CGM Use <sup>††</sup> | | | ~2 Week Blinded<br>CGM Use | Start of 26-Week<br>Unblinded CGM<br>Use | х | Х | Х | Х | х | |

<sup>\*</sup>Virtual Clinic Training and Follow up phase ends at 26 weeks. Participant will be asked to extend follow up for an additional 26 weeks and sign an addendum ICF if they plan to continue to use CGM after the first 26 weeks.

<sup>\*\*</sup>Participants will be asked to complete questionnaires monthly after CGM Initiation. A final questionnaire will be elicited at the earlier of CGM discontinuation or completion of study follow up (~52 weeks).

<sup>\*\*\*</sup>HbA1c checks prior to unblinded CGM initiation, and at 3-month intervals following CGM initiation (~13 weeks, 26 weeks, 39 weeks, and 52 weeks)

<sup>\*</sup>Follow up may be via phone, text, virtual (i.e. Skype), or app. outside of scheduled training. Additional follow up may be conducted as needed. Participants may follow up with study team as needed.

<sup>\*\*</sup>CGM supplied for blinded data collection will be provided. CGM supplies for six months of unblinded use will be provided for those who successfully complete blinded data collection.

## **3 Statistical Hypotheses**

- 2 There are no primary outcomes and additional analyses not pre-specified here may be performed.
- 3 In this study, we expect that most hypothesis testing will involve testing whether the change
- 4 from baseline for various outcomes is significantly different from zero. This will primarily be
- 5 for the CGM metrics, HbA1c, and the questionnaires. In those cases, the null hypothesis of the
- 6 change from baseline being equal to zero will be tested against the alternative hypothesis that the
- 7 change from baseline is nonzero. Analyses will be stratified by type of diabetes.

## 8 4 Sample Size

- 9 The goal for the study is to include at least 300 participants who initiate CGM. This is a
- 10 convenience sample and not based on statistical principles.

#### 5 Outcome Measures

- 12 The following quantitative study outcome measures will be tabulated by diabetes type using
- summary statistics appropriate to the distribution:
- HbA1c

11

19

20

26

27

29

30

32

33

34

36

37

- Percentage of time using the CGM
- Hours of CGM use
- Mean of sensor glucose levels
- Percentage of time spent with sensor glucose levels <54 and <70 mg/dL
  - Percentage of time spent with sensor glucose levels >180 and >250 mg/dL
  - Percentage of time spent with sensor glucose levels in the target range (70-180 mg/dL)
- Glycemic variability measured by the coefficient of variation
- Total daily insulin (units/kg)
- Total daily basal insulin (units/kg)
- Total daily bolus insulin (units/kg)
- Patient Health Questionnaire-8
  - Diabetes Distress Scale Management Distress Subscale
    - Hypoglycemia Fear Survey Worry Subscale
- CDC Healthy Days
  - Hypoglycemia Confidence Survey
    - Diabetes Technology Attitudes Survey
- Glucose Monitoring Satisfaction Survey
  - Openness Subscale
  - Emotional Burden Subscale
    - Behavioral Burden Subscale
- o Trust Subscale
  - Sleep Quality Scale
    - Benefits and Barriers of CGM Survey
- Percentage of CGM discontinuations
- CGM Discontinuation Survey (only administered to subjects who discontinue CGM)
- Positive screen for mental health

- o Positive screen triggered by Patient Health Questionnaire-8
  - o Positive screen triggered by Diabetes Distress Scale
    - o Positive screen triggered by Hypoglycemic Fear Survey Worry Scale
  - Behavioral health service utilization
    - Behavioral health metrics
    - Cost of care over time
    - Service utilization such as hospitalizations, ER visits, prescriptions filled

47 48

52

53 54

55

56

57

58

59

60

61 62

63

64

42

43

44

45

46

- 49 CGM, HbA1c, and insulin outcomes will be evaluated at baseline and 13, 26, 39, and 52 weeks.
- 50 CGM and insulin outcomes will also be evaluated over the first 26 weeks and last 26 weeks.
- Questionnaires will be evaluated at all time points they are collected.

# 6 Description of Statistical Methods

## **6.1** Analysis Cohorts

- All subjects enrolled in the study who initiate the CGM and have at least 168 hours of CGM data will be included in the tabulations of demographics and the glycemic outcome measures listed in Section 5
- CGM use assessment will include all subjects who stayed in the study at least one week following CGM initiation.
- HbA1c, questionnaires, insulin, and other analyses will include all subjects with any amount of corresponding data following CGM initiation.
- The tabulations of the safety outcomes will include all participants who enrolled, regardless of how much data is available.

# 7 Analysis of Study Endpoints

#### 7.1 Calculation of CGM Metrics

#### 7.1.1 Calculation of 13 Week CGM Metrics

- All CGM metrics listed in Section 5 will be calculated on a 13-week period for each subject
- level. The windows for the 13-week periods are defined as follows:

| Time Point | Window |
|-------------|-----------------------------------------------|
| 1-13 Weeks | 0 to 91 days after the CGM initiation date |
| 14-26 Weeks | 92 to 183 days after the CGM initiation date |
| 27-39 Weeks | 184 to 274 days after the CGM initiation date |
| 40-52 Weeks | 275 to 365 days after the CGM initiation date |

68

For each 13-week period, CGM metrics will be calculated by pooling all CGM readings

occurring from 12:00 AM on the first day of the 13-week period up until 11:59PM on the last

day of the 13-week period. For the first 13-week period, the first CGM reading will be the start

datetime of the period. If a participant discontinues CGM prior to the last day of the 13-week

period, then CGM data will include readings up to the last CGM reading on the discontinuation

date. Calibrations will be excluded from all these calculations. CGM metrics for 13-week periods

vith less than 168 hours of CGM data will be set to missing.

- 76 Baseline CGM metrics will be calculated by pooling all blinded CGM readings up to 90 days
- prior to the date of CGM initiation for each subject. Baseline CGM metrics with less than 72
- 78 hours of CGM data will be set to missing.
- 79 The amount of time using the CGM will be calculated as the number of CGM values multiplied
- by the expected CGM measurement frequency (i.e., 5min in general), with the exception that
- 81 there can only be one value within the CGM measurement frequency. Percentage of time CGM
- is used will be calculated as the amount of time using the CGM divided by the total possible time
- 83 the participant could have used the CGM during the same period. Note that this denominator
- includes sensor warm-up periods with no CGM values, so this metric will serve as a conservative
- estimate of CGM use.

#### 7.1.2 Calculation of 4 Week CGM Metrics

- 87 All CGM metrics listed in Section 5 also will be calculated on a 4-week interval for each subject.
- 88 The windows of the 4-week periods is defined as follows:

| Time Point | Window |
|-------------|-----------------------------------------------|
| 1-4 Weeks | 0 to 28 days after the CGM initiation date |
| 5-8 Weeks | 29 to 56 days after the CGM initiation date |
| 9-12 Weeks | 57 to 84 days after the CGM initiation date |
| 13-16 Weeks | 85 to 112 days after the CGM initiation date |
| 17-20 Weeks | 113 to 140 days after the CGM initiation date |
| 21-24 Weeks | 141 to 168 days after the CGM initiation date |
| 25-28 Weeks | 169 to 196 days after the CGM initiation date |
| 29-32 Weeks | 223 to 224 days after the CGM initiation date |
| 33-36 Weeks | 225 to 252 days after the CGM initiation date |
| 37-40 Weeks | 253 to 280 days after the CGM initiation date |
| 41-44 Weeks | 281 to 308 days after the CGM initiation date |
| 45-48 Weeks | 309 to 336 days after the CGM initiation date |
| 49-52 Weeks | 337 to 365 days after the CGM initiation date |

89

97

86

- 90 For each 4-week interval, CGM metrics will be calculated by pooling all CGM readings
- occurring from 12:00 AM on the first day of the 4-week interval up until 11:59PM on the last
- day of the 4-week period. For the first 4-week interval, the first day will be the day after CGM
- 93 initiation date. If a participant discontinues CGM prior to the last day of the 4-week period, then
- CGM data will include readings up to the day before CGM discontinuation date. Calibrations
- will be excluded from all these calculations. CGM metrics for 4-week periods with less than 168
- 96 hours of CGM data will be set to missing.

#### 7.1.3 Calculation of CGM Metrics during the First and Last 26 Weeks of the Study

- 98 All CGM metrics listed in Section 5 also will be calculated for the first and last 26 weeks of the
- 99 study for each subject. CGM metrics will be calculated by pooling all CGM readings in the first
- 26 weeks (i.e., 1-13 and 14-26 week periods defined above) and last 26 weeks (i.e., 27-39 and
- 40-52 week periods defined above). In these calculations, subjects that discontinue use of the
- 102 CGM during the period of time that is being evaluated will also be handled in the same way as

described above. Calibrations will be excluded from the calculations. CGM metrics for 26-week periods with less than 168 hours of CGM data will be set to missing.

#### 7.2 Calculation of Questionnaire Scores

Data from the following questionnaires will be reported at each time point collected:

- Patient Health Questionnaire-8: This questionnaire consists of 8 items, and it is typically used to screen for depression. Each item is scored on a scale of 0 to 3, with a higher value denoting more depressive symptoms. The total score is calculated by summing the individual responses to each question. Per the scoring instructions, total scores are set to missing for participants who skip more than one question. A total score of ≥10 denotes major depression, and a score of ≥20 denotes severe major depression.
- Diabetes Distress Scale Management Distress Subscale: This questionnaire consists of questions about the participant's distress regarding diabetes management. Items are ranked on a scale of 1 to 6, where a 1 denotes that the item is not a problem at all and a 6 denotes that it is a very serious problem. For this questionnaire, a mean score will be calculated across all questions.
- Hypoglycemia Fear Survey Worry Subscale: This questionnaire consists of items asking
  the participant about his or her worries regarding what may occur as a result of low blood
  sugar. Items are scored on a scale of 0 to 4. Higher numbers denote responses that are
  more worrisome. The total score is calculated by summing the responses to each
  question.
- CDC Healthy Days: This is a questionnaire about the participant's general mental and physical health. It estimates the number of days that the participant's mental and physical health has been adequate over the past month, in addition to the impact that the participant's health has had on his or her daily life. Analyses will report the percentage of participants ranking their general health as either fair or poor. Additionally, the number of unhealthy days over the past 30 days will be calculated by summing the number of reported unhealthy mental and physical days. The sum will be truncated at 30 days if it exceeds 30.
- Hypoglycemia Confidence Survey: This questionnaire asks the participant about their level of confidence regarding the avoidance of problems with daily activities due to hypoglycemia. Items are ranked on a scale of 1 to 4, with higher numbers denoting a higher level of confidence. For this questionnaire, a mean score will be calculated across questions.
- Diabetes Technology Attitudes Survey: This questionnaire consists of 5 questions about diabetes technology. Responses to each question are ranked on a scale of 1 to 5. Higher numbers denote more satisfaction with diabetes technology. A total score is calculated as the sum of the individual responses to each question.
- Glucose Monitoring Satisfaction Survey: This questionnaire asks the participant to provide a response on a scale of 1 to 5 to several questions about their satisfaction with their current glucose monitor. The directionality of the responses varies across questions, so some questions are reverse scored in the calculation of scores. The questionnaire includes four subscales, and the overall score is tabulated as a mean across all questions for the full questionnaire and each subscale.

- Sleep Quality Scale: This questionnaire consists of a single item asking the participant to rank their sleep quality on a scale of 0 to 10, with a higher number denoting better sleep. For this questionnaire, a mean score will be calculated across questions.
  - Benefit of CGM Survey: This questionnaire asks the participants questions about things that are good about wearing a CGM. The participants are asked to rank their agreement with each statement on a scale of 1 to 5. A higher number indicates more agreement, which would imply more satisfaction with using a CGM. For this questionnaire, a mean score will be calculated across questions.
  - Barriers of CGM Survey: This questionnaire asks the participants questions about things that are bad about wearing a CGM. The participants are asked to rank their agreement with each statement on a scale of 1 to 5. A higher number indicates more agreement, which would imply less satisfaction with using a CGM. For this questionnaire, a mean score will be calculated across questions.
  - CGM Discontinuation Survey (only administered to subjects who discontinue CGM): This questionnaire asks the participants several questions about why they discontinued CGM. For this survey, only responses to each individual question will be tabulated.

The electronic data capture system for this study will allow the subjects to skip questions on the questionnaires. For all questionnaires, at least 75% of questions must be answered in order to be included in the analyses (unless specified otherwise above). The 75% rule described above will be applied separately for the mean score and each subscale so it is possible that the sample size will be different for some subscales. The score used for the analyses will only be based on the questions that were answered. Analyses will be limited to subjects who are included in the primary cohort (no imputation).

#### **7.3 Missing Data**

146

147

148

149

150

151

152

153

154

155

156

157

158

159

160

161 162

163

164

165

166

167

168

169

- 171 Missing data will not be imputed for any outcomes in this study and will be handled by means of
- direct likelihood analyses.

#### 173 7.4 Statistical Methods

- For all outcomes, summary statistics appropriate to the distribution will be tabulated on a subject
- level overall and within the subgroups defined in Section 12. For the CGM metrics, summary
- statistics appropriate to the distribution also will be tabulated for each 4-week interval and for the
- first and last 26 weeks of the study. For the questionnaires, summary statistics will be reported
- for the mean scores in addition to the individual responses for each question.
- 179 For all outcomes, a linear mixed model with a random subject effect will be used to test whether
- the mean change from baseline significantly differs from zero. These models will be fit for each
- of the subject level CGM metrics and HbA1c at 13, 26, 39, and 52 weeks. They also will be fit
- for the questionnaires at 26 and 52 weeks. If values are skewed, then winsorization will be
- utilized. Point estimates and 95% confidence intervals for change in glycemic outcomes will be
- 184 reported.
- For the three mental health screening questionnaires, only summary statistics will be tabulated.
- The three mental health screening questionnaires falling under this umbrella are the Patient

- Health Questionnaire-8, the Diabetes Distress Scale (Management Distress Subscale), and the
- 188 Fear of Hypoglycemia Survey (Worry Subscale).

#### 189 7.5 Analyses Windows

- 190 For HbA1c, only measurements occurring within ±45 days of the target measurement date at a
- 191 given time point will be included in the tabulation of summary statistics. The windows for
- 192 glycemic metrics were defined above in Section 7.1.

#### 193 **7.6 Sensitivity Analyses**

- 194 For CGM and HbA1c outcomes, a complete-case analysis restricting to non-missing outcomes
- will also be assessed. A paired t-test (for normally distributed outcomes) or a Wilcoxon signed
- rank test (for skewed outcomes) will be used.

## 197 8 Safety Analyses

- All adverse events that occur on or after the date of enrollment will be listed in a table.
- 199 For events occurring on or after the date of CGM initiation, the reported safety outcomes include
- diabetic ketoacidosis (DKA), severe hypoglycemia (SH), hospitalization, and emergency room
- visits. The following statistics will be tabulated for each safety outcome:
- Total number of events

203

205

209

- Number and proportion of subjects with an event (discretized into bins)
- Incidence rate per 100 person years
- The number of person-years for the incidence rate calculations will be inclusively defined as the
- 207 number of person-years in between the CGM initiation date and the last day of study follow-up
- 208 (completion date, withdrawal date, etc.).

# 9 Adherence and Retention Analyses

#### 210 9.1 Protocol Adherence

- The number of and reasons for participant contacts with the virtual clinic will be reported in a
- table to assess protocol adherence for the study.

# 213 10 Baseline Descriptive Statistics

- Baseline demographic and clinical characteristics of the cohort of all subjects who initiate the
- 215 CGM and were included in the glycemic analyses will be summarized in a table. Use of
- 216 medications and non-insulin therapy will also be reported. For continuous variables, summary
- statistics appropriate to the distribution will be given. For discrete variables, number and
- 218 percentage will be reported for each category. Summary statistics for demographics and clinical
- 219 characteristics will be presented overall, by diabetes type, by insulin modality, by whether the
- participant was seeing an endocrinologist or a primary care provider at baseline, by baseline
- 221 HbA1c groups (<7.5%, 7.5% to <9.0%, and  $\ge9.0\%$ ), and by age (<25, 25-65, and >65 years). Cut
- points for age and baseline HbA1c may be reassessed after data are collected.

## 223 11 Planned Interim Analyses

- No formal interim analyses or stopping guidelines are planned for this study. Data will be
- 225 monitored on an ongoing basis including:
- Status of enrolled participants
- Recruitment rates by month and by site
- Baseline demographic and clinical characteristics
- Dropped participants and reasons for discontinuing
- Reportable adverse events

## 12 Subgroup Analyses

- Subgroup analyses for % of time using the CGM, % time in range, % time >180 mg/dL, % time
- 233 <70 mg/dL, and HbA1c will be performed based on the following factors:
- Baseline HbA1c (categorized as <7.5%, 7.5% to <9.0%, and ≥9.0%)
- Insulin modality

231

- Age (categorized as <25, 25-65, and >65)
- Type of healthcare provider (endocrinologist or primary care provider)
- Diabetes Duration (categorized as <5, 5-<10, 10-<20, ≥20)
- Race/Ethnicity
- Household income (categorized as <\$50,000, \$50,000-<\$100,000, and ≥\$100,000)
- 241 For continuous variables, results will be displayed in subgroups based on cut points although the
- analysis will utilize the variable as continuous. Cut points for age, baseline HbA1c, diabetes
- 243 duration, and household income may be reassessed after the data are collected.
- Within each subgroup, summary statistics will be tabulated. P-values for change from baseline
- 245 will be calculated within each subgroup using a linear mixed model will be performed as
- described in Section 7.4.
- 247 Percentage of CGM discontinuations will also be tabulated by the factors listed above.

# 248 13 Multiple Comparisons

No adjustments for multiple comparisons will be made.

# 250 14 Additional Analyses

- 251 CGM metrics over 13-week periods will be tabulated on a subject level by time of day. In these
- analyses, daytime will be defined as 6:00 AM to <12:00 AM and nighttime will be defined as
- 253 12:00 AM to <6:00 AM. For this analysis, CGM metrics will only be calculated if the participant
- has at least 126 hours of CGM data during daytime and at least 42 hours of CGM data during
- 255 nighttime.
- Total scores for questionnaires in Section 7.2 will be stratified by number of mental health
- service sessions. Additional analyses will be conducted to assess the bivariate relationship
- between questionnaire responses and glycemic metrics at 26 and 52 weeks. These relationships
- will be assessed by displaying scatterplots, along with the corresponding Spearman correlation

- coefficient. A 95% confidence interval for the Spearman correlation coefficient will be reported.
- In these analyses, the following relationships will be explored:

263

264

- % Time <70 mg/dL vs. Fear of Hypoglycemia Worry Subscale Mean Score
  - % Time <70 mg/dL vs. Hypoglycemia Confidence Survey Mean Score
  - % Time in Range vs. Glucose Monitoring Satisfaction Survey Mean Score
- % Time in Range vs. Diabetes Distress Scale Management Distress Subscale Mean Score
- CGM use at 26 weeks vs. Diabetes Technology Attitudes Survey Mean Score